CLINICAL TRIAL: NCT03067519
Title: Fast Track Surgery for Abdominal Surgery in Rwanda: a Randomized Controlled Trial
Brief Title: Fast Track Surgery for Abdominal Surgery in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rwanda (Other)
Responsible Party: Principal Investigator, Ndayizeye Leonard, consultant surgeon, honorary lecturer university of Rwanda, University of Rwanda
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URwanda
Record Dates: First submitted 2017-02-21; First posted 2017-03-01 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Elective Surgical Procedures

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients were randomly put in group using sealed envelop.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast track surgery (Experimental): Intervention: Fast track surgery patients underwent early feeding and mobilization after surgery
  Interventions: Other: Fast track surgery
- Conventional management (Active Comparator): usual postoperative care per surgeon
  Interventions: Other: Conventional management

INTERVENTIONS:
Other: Fast track surgery — early feeding and mobilization after surgery
  Arms: Fast track surgery
Other: Conventional management — Management per the primary surgeon
  Arms: Conventional management

SUMMARY:
Fast Track Surgery (FTS) was started in colorectal surgery, but was later applied to other surgical fields. Core elements include epidural or regional anaesthesia, perioperative fluid management, minimally invasive surgical techniques, pain control, and early mobilization and feeding. Beneficial effects of FTS include reduced costs, early hospital discharge, and increased availability of hospital beds.The main aim of this study was to explore the efficacy of FTS in the Rwandan surgical setting and to demonstrate the benefits of FTS.

it is study comparing the management of surgical patients using traditional management and fast track surgery. the study was done on patients undergoing elective abdominal surgery only

DETAILED DESCRIPTION:
Fast track surgery (FTS) uses a multifaceted approach to reduce the stress response to surgery, thereby improving outcomes and decreasing length of hospital stay. The core elements of FTS include: epidural or regional anesthesia, peri-operative fluid management, minimally invasive techniques, optimal pain control, early initiation of oral feeding and early mobilization. The combination of these approaches has led to a significant reduction in complication rates, morbidity and mortality rates, duration of hospital stay and costs of hospitalization, and greatly improved postoperative recovery The main aim of this study was to explore the efficacy of FTS in the Rwandan surgical setting and to demonstrate the benefits of FTS.

This randomized control trial was conducted in CHUK over a period of three months (October - December, 2015). For patients in the FTS arm, the study investigator would assess patients on a daily basis and work with the primary surgical team. The study investigator would prompt the primary surgical team for early feeding, mobilization, pain control and fluid management recommendations.

Data were collected on variables including postoperative analgesia, mobilisation, resuming oral feeding, hospital stay and complications. The primary outcome was duration of postoperative hospital stay and secondary outcome was major complications.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted for elective abdominal surgery

Exclusion Criteria:

* patients with comorbidity, American Society of Anesthesiologists score greater than 2

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
hospital stay | within 30 days
  numbers of days spent in hospital

SECONDARY OUTCOMES:
Major complications | within 30 days
  Major complications were defined as: in-hospital death, intra-abdominal abscess, anastomotic leak, surgical site infection, pneumonia, urinary tract infection, and venous thromboembolism.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED KISWEZI, MMed, Study Director — University of Rwanda
Locations (1):
- university teaching hospital Kigali, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No